CLINICAL TRIAL: NCT05720637
Title: The Efficacy and Cerebral Mechanism of Intradermal Acupuncture for Major Depressive Disorder: a Study Protocol for a Randomized Controlled Trial
Brief Title: The Efficacy and Cerebral Mechanism of Intradermal Acupuncture for Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaomei Shao (Other)
Collaborators: Zhejiang Provincial Tongde Hospital (Other); First People's Hospital of Hangzhou (Other); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor-Investigator, Xiaomei Shao, Professor, The Third Affiliated hospital of Zhejiang Chinese Medical University
Organization: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022ZX010-IAM
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Intradermal Acupuncture; Magnetic Resonance Imaging
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Waiting list group (Other): This group will include 40 patients with MDD who will be treated with oral SSRIs only, the dosage of which will be determined by the psychiatrist. At the end of this trial, patients could choose 6 weeks' intradermal acupuncture treatments free of charge.
  Interventions: Drug: SSRI
- SIA group (Sham Comparator): This group will include 40 patients with MDD who will be treated with sham intradermal acupuncture (SIA) combined with SSRIs. Acupoints related to MDD will be stimulated by acupuncturists and the dosage of oral SSRIs will be determined by the psychiatrist.
  Interventions: Drug: SSRI; Device: SIA
- AIA group (Experimental): This group will include 40 patients with MDD who will be treated with active intradermal acupuncture (AIA) combined with SSRIs. Acupoints related to MDD will be stimulated by acupuncturists and the dosage of oral SSRIs will be determined by the psychiatrist.
  Interventions: Drug: SSRI; Device: AIA

INTERVENTIONS:
Drug: SSRI — SSRIs antidepressants, including fluoxetine, paroxetine, sertraline, citalopram, etc., will be administered at oral doses determined by the psychiatrist. Once daily for the duration of the trial.
  Other Names: selective 5-hydroxytryptamine reuptake inhibitor
Device: SIA — This study will select 4 acupoints (all taken bilaterally) commonly used to treat MDD, namely Taichong (LR3), Neiguan (PC6), Sanyinjiao (SP6) and Shenmen (HT7). The SIA will use the same size, colour and material as the AIA with a thin silicone pad in the middle instead of the needle body. SIA will be attached to the acupoints and retained for 72 hours, removed and rested for one day. A total of 10 sessions will be performed over a period of 6 weeks.
  Other Names: sham intradermal acupuncture
  Arms: SIA group
Device: AIA — This study will select 4 acupoints (all taken bilaterally) commonly used to treat MDD, namely Taichong (LR3), Neiguan (PC6), Sanyinjiao (SP6) and Shenmen (HT7). Depending on acupoints' location, a φ0.20*1.5mm or φ0.20*1.2mm AIA will be selected. Press the AIA to insert it vertically into the acupoint and retain it in the skin. AIA will be retained for 72 hours with a day's rest after removal. During the period of needle retention, participants will be instructed to press the AIA 3-4 times a day for approximately 1 minute each time, with as much stimulation as the patient can tolerate, at intervals of approximately 4 hours. A total of 10 sessions will be performed over a period of 6 weeks.
  Other Names: active intradermal acupuncture
  Arms: AIA group

SUMMARY:
Major depressive disorder (MDD) is highly prevalent, affecting nearly 4% of the global population. Pharmacotherapy is the frontline treatment recommended by the guideline, but it also has some limitations such as delayed onset, inadequate response, and drug resistance. Intradermal acupuncture (IA) is a method of using short indwelling needles retained under the skin to produce continuous stimulation for long-term efficacy. It has been reported that IA combination medication appears to be more valuable than medication alone in the treatment of MDD, however, there is a lack of high-quality clinical evidence.While several studies have proposed that manual or electroacupuncture can improve MDD symptoms by modulating brain networks, the cerebral mechanism of IA as superficial acupuncture for MDD has not been reported. Hence, investigators designed a multicentre randomized controlled trial to assess the clinical efficacy and safety of IA for MDD and preliminarily explore the potential therapeutic mechanisms for IA by functional magnetic resonance imaging (fMRI) .

DETAILED DESCRIPTION:
A total of 120 patients with MDD who meet the inclusion criteria will be included in the study. Participants will be randomly assigned 1:1:1 to the waiting list group (patients in this group will be treated with selective 5-hydroxytryptamine reuptake inhibitors (SSRIs) only), sham intradermal acupuncture combined with SSRIs (SIA) group and active intradermal acupuncture combined with SSRIs (AIA) group. The study will assess the efficacy and safety of intradermal acupuncture for MDD. In addition, investigator will explore the possible cerebral mechanisms by which IA exerts its antidepressant effects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with MDD according to the International Classification of Disease-10 (ICD-10);
2. Aged between 18 and 60 years (no limitation on gender);
3. Administration of SSRIs;
4. Patients undergoing MRI and MRS should be right-handed and free of traumatic brain injury, claustrophobia or metal implants;
5. Written informed consent is obtained by the person or guardian.

Exclusion Criteria:

1. ICD-10 diagnoses: schizophrenia, bipolar disorder, manic episode or other psychotic disorders; alcohol and drug addiction;
2. Significant skin lesions, severe allergic diseases, tumors, and severe or unstable internal diseases involving the cardiovascular, digestive, endocrine, or hematological system;
3. Acute suicidal tendency;
4. Allergy to adhesive tape and fear of intradermal acupuncture;
5. Pregnancy and lactation;
6. Mental retardation and difficulty cooperating with doctors.
7. Participating in other clinical trials.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Changes in the Hamilton Depression Scale-17 (HAMD-17) Scores | Baseline, 3 weeks after treatment, 6 weeks after treatment, at 4-week follow-up.
  The HAMD scale is the most commonly used in the clinical assessment of depression, including 17 items. The higher the score, the more severe the depression. 0-7 means no depressive symptoms, 8-17 means mild depression, 18-24 was divided into moderate depression, and 25-52 was divided into severe depression.

SECONDARY OUTCOMES:
Changes in the Self-Rating Depression Scale (SDS) Scores | Baseline, 3 weeks after treatment, 6 weeks after treatment, at 4-week follow-up.
  The standard score is the total of all scores multiplied by 1.25 to the nearest whole number on this scale, which has 20 questions. A standard score below 50 is normal; 50-60 is mild depression; 61-70 is moderate depression; 70 or more is severe depression.
Changes in the Pittsburgh Sleep Quality Index (PSQI) Scores | Baseline, 3 weeks after treatment, 6 weeks after treatment, at 4-week follow-up
  The PSQI is used to assess the sleep quality of the participant in the last 1 month and consisted of 19 self-rated and 5 other rated items. The higher the score, the worse the sleep quality. Sleep quality is divided into 4 levels according to the total score.

OTHER OUTCOMES:
Magnetic resonance imaging (MRI) data acquisition | Baseline
  Brain MRI will be taken by a 3.0T MRI scanner to analyze the activity function of brain regions, such as the striatum and ventral tegmental area, before and after the acupuncture intervention of patients, and at the baseline of heath controls.
Evaluation of acupuncture compliance | 6 weeks after treatment
  At the end of the acupuncture intervention (end of week 6), compliance will be evaluated with the formula: Compliance Rate = (actual treatment times/total treatment times) *100%.
Adverse Events | Up to 10 weeks
  Adverse events such as bleeding, haematoma, or unbearable pain caused by the needle, as well as drug-induced nausea, vomiting or dizziness, will all be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomei Shao, Ph.D, Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University
Locations (1):
- the Third affiliated hospital of Zhejiang Chinese Medical university [Recruiting], Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Wu X, Tu M, Chen N, Yang J, Jin J, Qu S, Xiong S, Cao Z, Xu M, Pei S, Hu H, Ge Y, Fang J, Shao X. The efficacy and cerebral mechanism of intradermal acupuncture for major depressive disorder: a study protocol for a randomized controlled trial. Front Psychiatry. 2023 May 15;14:1181947. doi: 10.3389/fpsyt.2023.1181947. eCollection 2023. PMID 37255689